CLINICAL TRIAL: NCT04792606
Title: Long-Term Outcomes of Hip Interventions for Children With Cerebral Palsy - An International Multi-Centre Prospective Comparative Cohort Study (CHOP-II)
Brief Title: Long-Term Outcomes of Hip Interventions for Children With Cerebral Palsy
Acronym: CHOP II
Status: Recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Royal Children's Hospital (Other); Shriners Hospitals for Children,Canada (Unknown); Provincial Health Services Authority British Columbia (Other); Aarhus University Hospital (Other); Sheba Medical Center (Other Government); Seoul National University Bundang Hospital (Other); Starship Children's Hospital of New Zealand (Unknown); Poznan University of Medical Sciences (Other); Skane University Hospital (Other); Karolinska University Hospital (Other); Great Ormond Street Hospital for Children NHS Foundation Trust (Other); The Royal London Hospital (Unknown); Nuffield Orthopaedic Centre NHS Trust (Other); Children's Hospital Medical Center, Cincinnati (Other); Boston Children's Hospital (Other); Columbia University (Other); Shriners Hospitals for Children, Sacramento (Unknown); Gillette Children's Specialty Healthcare (Other); Alfred I. duPont Hospital for Children (Other); IWK Health Centre (Other); Alder Hey Children's NHS Foundation Trust (Other); Children's Hospital Colorado (Other); Hospital for Special Surgery, New York (Other); Shriners Hospitals for Children, Honolulu (Unknown); Robert Jones and Agnes Hunt Orthopaedic and District NHS Trust (Other Government); Morgan Stanley Children's Hospital (Other); Children's Health Queensland Hospital and Health Service (Unknown); University of Nebraska (Other)
Responsible Party: Principal Investigator, Unni Narayanan, MBBS, MSc, FRSC(C), The Hospital for Sick Children
Other Study IDs: 420492
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy
Keywords: non-ambulatory, non-ambulatory cerebral palsy, patient reported outcomes measures, PROMS, outcomes, CPCHILD
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- "Natural" History or watchful waiting
- Serial botulinum toxin injections
- Adductor (+/- psoas) muscle releases alone
- Hip reconstructive surgery
- Salvage hip surgery

SUMMARY:
Children with severe cerebral palsy (CP) are at high risk for progressive hip displacement, associated with pain and contractures interfering with many aspects of care, comfort and quality of life. These children undergo many types of interventions, the optimal timing and effectiveness of which, remain unclear. In 2014, CIHR funded the CP Hip Outcomes Project (CHOP), an international multi-centre prospective longitudinal cohort study of children with severe (non-ambulant) CP with evidence of hip displacement defined as a Reimer's migration percentage (MP) of at least 30%. The study was designed to evaluate the comparative effectiveness of different treatment strategies to prevent or relieve symptoms associated with hip instability, using the validated Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD ) questionnaire as the primary outcome measure of health-related quality of life © (HRQL) for this population. 650 patients enrolled from 28 sites in 11 countries, are actively being followed and will reach at least 2 years of follow-up at the end of 2019. This project, will study the impact of hip instability and its management in children with severe CP using the CPCHILD questionnaire that was developed specifically for this purpose. Although CHOP will define outcomes at 24 months, the outcomes are not expected to remain stable while the child is still growing. The inception cohort will need follow-up until skeletal maturity to track their long-term outcome trajectories.

DETAILED DESCRIPTION:
Background: Children with severe cerebral palsy (CP) are at high risk for progressive hip displacement, associated with pain and contractures interfering with many aspects of care, comfort and quality of life. These children undergo many types of interventions, the optimal timing and effectiveness of which, remain unclear. In 2014, CIHR funded the CP Hip Outcomes Project (CHOP), an international multi-centre prospective longitudinal cohort study of children with severe (non-ambulant) CP with evidence of hip displacement defined as a Reimer's migration percentage (MP) of at least 30%. The study was designed to evaluate the comparative effectiveness of different treatment strategies to prevent or relieve symptoms associated with hip instability, using the validated Caregiver Priorities and Child Health Index of Life with Disabilities (CPCHILD ) questionnaire as the primary outcome measure of health-related quality of life © (HRQL) for this population. 650 patients enrolled from 28 sites in 11 countries, are actively being followed and will reach at least 2 years of follow-up at the end of 2019. This project, unique in scale and design, will study the impact of hip instability and its management in children with severe CP using a meaningful outcome measure that was developed specifically for this purpose. Although CHOP will define outcomes at 24 months, the outcomes are not expected to remain stable while the child is still growing. The inception cohort will need follow-up until skeletal maturity to track their long-term outcome trajectories. The international network of investigators/sites and the infrastructure established for CHOP will facilitate the long-term follow-up of the participants in this study. In addition, the results of CHOP will inform the design of nested trials to evaluate the effectiveness of future interventions aimed at improving the quality of life of children with severe disabilities.

Study Aims Aim 1: Measure the post 24-month effectiveness of different treatment strategies for hip displacement in children with severe CP using the CPCHILD as the primary outcome measure.

Aim 2: Compare the rates of recurrence, relapse of symptoms, additional interventions and other longer term complications associated with each of the treatment cohorts.

Methods

Study Design: Multi-centre longitudinal cohort study of children with severe (non-ambulant) CP, ages 3 to 18 years with hip MP ≥ 30% enrolled in one of 5 cohorts:

A. "Natural" History or watchful waiting B. Serial botulinum toxin injections C. Adductor (+/- psoas) muscle releases alone D. Hip reconstructive surgery E. Salvage hip surgery Data collected include demographics, prognostic factors, including co-morbid conditions, parental reports of HRQL as measured by the CPCHILD, and radiographic measures of MP and acetabular index (AI). The primary outcome measure CPCHILD, as well as the MP & AI will be assessed every 12 months after the 24 month follow-up since inception in CHOP. The cohort of 650 children enrolled in Groups B, C, D, & E will be compared with each other as well as with their respective propensity matched counterparts of untreated children (Group A), using repeated measures ANOCOVA at 3yrs, and annually thereafter until at least 5 years of follow-up or skeletal maturity.

Significance: CHOP I & II will establish the superiority of either prophylactic or reactive intervention strategies for hip displacement in severe CP and provide justification for hip surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Children with severe, non-ambulant (GMFCS IV & V) Cerebral Palsy
* between 2 and 19 years of age
* with radiographic evidence of hip displacement (previously untreated) as measured by Reimer's MP ≥ 30%
* and their parents or primary caregivers, defined as the individual most involved in the daily care of the child are willing to complete the CPCHILD in one of the available languages the CPCHILD is offered in

Exclusion Criteria:

* under the age of 2, or over the age of 19
* Reimer's migration percentage under 30% in both hips
* parents or primary caregivers unable to complete the CPCHILD in one of it's available languages

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children between the ages of 2 and 19 with severe cerebral palsy (defined as a GMFCS level or IV or V) experiencing hip displacement (with radiographic evidence of a migration percentage (MP) or 30%) will be recruited to be apart of the CHOP II study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Caregiver Priorities & Child Health Index of Life with Disabilities (CPCHILD) | The CPCHILD takes approximately 15 minutes to complete
  The CPCHILD questionnaire is intended for persons with CP who rely on a wheelchair for most of their mobility. The CPCHILD questionnaire assesses how parents or caregivers rate their child (or how a child rates him/herself when able) about various issues related to daily activities, self care, getting around, comfort, communication, social interaction and health. The CPCHILD also identifies which of these issues the parents (or the child) feel are important to improve.

CONTACTS AND LOCATIONS:
Overall Officials: Unni G Narayanan, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No